CLINICAL TRIAL: NCT01763723
Title: Pigment-Tan-Safety Study of a Light-based Home Device for Hair Removal in Adult Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Christina Haak, MD., Bispebjerg Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: H-1-2012-025
Record Dates: First submitted 2012-12-20; First posted 2013-01-09 (Estimated); Last update posted 2015-07-31 (Estimated); Status verified 2015-07

CONDITIONS: Healthy
Keywords: Intense pulsed light,; UV-exposure,; skin type,; safety,; pigment,; home-use; subjects

ARMS (1):
- IPL after UV-exposure (Experimental): 8 UV-exposures followed by 3 weekly IPL exposures
  Interventions: Device: IPL-home use device

INTERVENTIONS:
Device: IPL-home use device — A light based home use device for hair removal

SUMMARY:
This studies was designed to investigate the importance of skin type and UV-exposure on side effects after exposure to an Intense Pulsed Light Home-use device.

21 healthy subjects will receive 8 UV-exposures on one buttock and subsequently three weekly IPL-exposures.

DETAILED DESCRIPTION:
Twenty-one healthy subjects will be exposed to UV-exposures 8 times over 3 weeks on a test-area (4 x 6cm) on one buttock to induce pigmentation. This will be followed by 3 weekly IPL (intense pulsed light) exposures. At 24 hours after the first IPL exposure, biopsies will be excised from the buttocks of the subjects (4 each).The skin will be evaluated after IPL exposure for: skin reactions, pain and mRNA expression of two pigment markers. Follow-up visits is planned at 1 and 4 weeks after the third and final IPL exposure.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, over 18 years, no childbearing potential, signed informed consent, no moles,tattoos, freckles or scars in the test-area, skin type II-IV

Exclusion Criteria:

* disease in test-area, prior treatment to IPL, taking drugs interfering with the immune system

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2012-04; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Changes in skin reaction development | Immediately after, 1 hr after, 16-24 hrs after, 1 week and 4 weeks after IPL exposure
  Redness, edema, pigment changes, texture changes, blisters and crusting

SECONDARY OUTCOMES:
Pain | Immediately after IPL exposure (approx. 2 min)

OTHER OUTCOMES:
mRNA expression of pigment markers | 16-24 hrs after the first IPL exposure

CONTACTS AND LOCATIONS:
Locations (1):
- Bispebjerg Hospital, Copenhagen, Bispebjerg, Denmark